CLINICAL TRIAL: NCT00595231
Title: A Multi-Center,Randomized, Double-Blind, Placebo-Controlled, Phase 2, Exploratory Study to Evaluate the Effect of Rufinamide on Anxiety in Patients With Moderate to Severe Generalized Anxiety Disorder
Brief Title: Exploratory Study to Evaluate the Effect of SYN111 (Rufinamide) in Patients With Generalized Anxiety Disorder (GAD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biotie Therapies Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYN111-CL03
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Generalized Anxiety Disorder
Keywords: GAD
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — rufinamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SYN111 (Experimental): 500 mg 1 week, followed by 1000 mg for 7 weeks
  Interventions: Drug: SYN111
- Placebo (Placebo Comparator): 0 mg tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYN111 — 500 mg for 1 week followed by 1000 mg for 7 weeks
  Other Names: Rufinamide
  Arms: SYN111
Drug: Placebo — 0 mg tablets
  Arms: Placebo

SUMMARY:
A Multi-Centered Randomized, Double-Blind, Placebo-Controlled, Phase 2, Exploratory Study to Evaluate the Effect of Rufinamide on Anxiety in Patients with Moderate to Severe Generalized Anxiety Disorder.

DETAILED DESCRIPTION:
This was an exploratory study to evaluate the effect of 500 or 1000 mg per day for 8 weeks of Rufinamide compared to placebo on measures of anxiety in patients with Generalized Anxiety Disorder, and to determine tolerability of Rufinamide in this population.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient 18-65
* Meet Diagnostic and Statistical Manual,(DSM) IV criteria for GAD
* Have moderate to severe anxiety
* Sign IRB (Institutional Review Board) approved consent and can comply with visits and procedures
* Women of childbearing potential must use acceptable method of contraception

Exclusion Criteria:

* Have diagnosis of adjustment disorder or anxiety disorder Not otherwise specified (NOS)
* Have diagnosis of specific phobia
* Have diagnosis of antisocial personality disorder or other Axis II Disorder
* Have diagnosis of substance abuse disorder within 3 months of study entry
* Have diagnosis of major depressive disorder or panic disorder within 6 months of study entry
* Have diagnosis of PTSD, eating disorder substance dependence disorder within 12 months of study entry
* Have diagnosis anytime during lifetime of schizophrenia or other psychotic disorder, bipolar mood disorder, Obsessive-Compulsive Disorder (OCD), psychosurgery
* Require medication to treat GAD other than study medication
* Failed to show improvement with past treatment for GAD
* Excessively consume caffeine
* Are receiving treatment with prohibited medications
* Uncontrolled thyroid condition
* Positive urine drug screen
* Obese
* Clinically significant ECG finding
* Participating in other clinical trial
* Clinically significant out of range lab value
* Past exposure to rufinamide
* Pregnant or nursing females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christpher Kenney, MD, Study Chair — Biotie Therapies Inc.
Locations (2):
- United States (2):
  - Carmen Research, Atlanta, Georgia
  - Midwest Clinical Research Center, Dayton, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 239 subjects were randomized into the trial from 19 of the 20 study sites initiated.
Groups:
- Rufinamide: 500 mg 1 week, followed by 1000 mg for 7 weeks
- Placebo: 0 mg. tablet
Period: Overall Study
Arm/Group | Rufinamide | Placebo
Started | 120 | 119
Completed | 115 | 114
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Population: ITT Population: Randomized and received at least one dose of the study drugs.
Groups:
- Rufinamide: 500 mg for 1 week followed by 1000 mg for 7 weeks
- Placebo: Placebo, 0 mg tablets
- Total: Total of all reporting groups
Arm/Group | Rufinamide | Placebo | Total
Number analyzed (Participants) | 115 | 114 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (12.47) | 35.6 (11.53) | 37.0 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 81 | 157
  Male | 39 | 33 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 19 | 31
  Not Hispanic or Latino | 103 | 95 | 198
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 12 | 8 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 14 | 17 | 31
  White | 82 | 69 | 151
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 18 | 25
Region of Enrollment [Number; unit: participants]
  United States | 115 | 114 | 229

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAMA) - Total Score: Summary Statistics - Observed
Description: The Hamilton Anxiety Scale is a 14-item test measuring the severity of anxiety symptoms. It provides measures of overall anxiety, psychic anxiety (mental agitation and psychological distress), and somatic anxiety (physical complaints related to anxiety). The interviewer then rated the individuals on a 5-point scale for each of the 14 items. Seven of the items specifically address psychic anxiety and the remaining 7 items address somatic anxiety. The total anxiety score ranges from 0 to 56. The 7 psychic anxiety items elicit a psychic anxiety score that ranges from 0 to 28. The remaining 7 items yield a somatic anxiety score that also ranges from 0 to 28. A score of 17 or less indicates mild anxiety severity. A score from 18 to 24 indicates mild to moderate anxiety severity, a score of 25 to 30 indicates a moderate to severe anxiety and lastly a score of 31-56 is very severe. HAM-A total score is the sum of items 1 - 14.
Time Frame: 8 Weeks
Population: ITT Population: Randomized and received at least one dose of the study drugs.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rufinamide | Placebo
Number analyzed (Participants) | 115 | 114
score on a scale
  Screening | 25.5 (3.70) | 25.6 (3.77)
  Baseline | 25.5 (3.77) | 25.8 (3.74)
  Week 1: number analyzed (Participants) | 114 | 114
  Week 1 | 21.9 (6.04) | 21.4 (5.71)
  Week 2: number analyzed (Participants) | 105 | 107
  Week 2 | 20.0 (6.29) | 19.6 (5.97)
  Week 3: number analyzed (Participants) | 102 | 101
  Week 3 | 18.0 (7.45) | 17.8 (7.02)
  Week 6: number analyzed (Participants) | 91 | 98
  Week 6 | 15.7 (7.34) | 16.7 (7.32)
  Week 8: number analyzed (Participants) | 84 | 92
  Week 8 | 15.1 (7.76) | 15.1 (7.19)
  Last Observation: number analyzed (Participants) | 114 | 114
  Last Observation | 16.7 (7.91) | 16.1 (7.65)

2. Primary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS). Summary Statistics
Description: The Hospital Anxiety and Depression Scale is a self screening questionnaire for depression and anxiety. It consists of 14 questions, seven for anxiety and seven for depression. The 14 statements are relevant to either generalized anxiety (7 statements) or 'depression' (again 7). Each question has 4 possible responses. Responses are scored on a scale from 3 to 0. The maximum score is therefore 21 for depression and 21 for anxiety. A score of 11 or higher indicates the probable presence of the mood disorder with a score of 8 to 10 being just suggestive of the presence of the respective state. The 2 subscales, anxiety and depression, have been found to be independent measures. In its current form the HADS is now divided into 4 ranges: normal (0-7), mild (8-10), moderate (11-15) and severe (16-21). Anxiety score = sum of items 1, 3, 5, 7, 9, 11, and 13. Depression score = sum of items 2, 4, 6, 8, 10, 12, and 14.
Time Frame: 8 Weeks
Population: ITT Population: Randomized and received at least one dose of the study drugs.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rufinamide | Placebo
Number analyzed (Participants) | 115 | 114
score on a scale
  Week 1 | -0.2 (2.66) | -0.1 (2.02)
  Week 2 | -0.4 (2.42) | -0.4 (2.69)
  Week 3 | -1.0 (3.14) | -0.5 (2.91)
  Week 6 | -1.4 (3.57) | -1.2 (3.20)
  Week 8 | -2.0 (3.61) | -1.6 (3.07)
  Last Observation | -1.2 (3.74) | -1.4 (3.01)

3. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Scale (MADRS) Summary Statistics.
Description: The MADRS (Montgomery and Asberg 1979) is a clinician-rated instrument that measures the presence and severity of depression. This instrument consists of 10 items. Each item is rated on a defined step scale of 0 to 6 with anchors at 2-point intervals. The MADRS total score is the sum of the 10 items and ranges from 0 to 60. A high numeric rating shows a greater degree of symptom severity.
Time Frame: 8 Weeks
Population: ITT Population: Randomized and received at least one dose of the study drugs.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rufinamide | Placebo
Number analyzed (Participants) | 115 | 114
score on a scale | 15.7 (5.51) | 16.4 (4.86)

4. Primary Outcome: Change From Baseline in Clinical Global Impression Scale for Severity of Illness: (CGI-S)
Description: Severity of illness is the first scale in the CGI. A rating is filled in by the investigator at the start of treatment based on a 0-7 point weighted scale. It goes from not assessed (0), to among the most extremely ill patients (7).
Time Frame: 8 weeks
Population: ITT Population: Randomized and received at least one dose of the study drugs.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rufinamide | Placebo
Number analyzed (Participants) | 115 | 114
score on a scale | 4.5 (0.60) | 4.4 (0.56)

5. Primary Outcome: Change From Baseline Raskin Depression Scale.
Description: It explores the extent to which an individual demonstrates depression on three sub-scales (rated 1-5): verbal self-report, behavior and secondary symptoms of depression. Scores range from 3-15, with higher scores indicating greater severity.
Time Frame: 8 weeks
Population: ITT Population: Randomized and received at least one dose of the study drugs.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rufinamide | Placebo
Number analyzed (Participants) | 115 | 114
score on a scale | 5.2 (1.22) | 5.3 (1.20)

6. Primary Outcome: Change From Baseline in Covi Anxiety Scale (CAS) - Index Total Score: Summary Statistics Observed
Description: The Covi Anxiety Scale is a simple 3 item scale for the assessment of severity of anxiety symptoms. The scale measures 3 dimensions: verbal report, behavior and somatic symptoms of anxiety. Each item scored on a scale of 1 - 5. (1)not at all, (2)somewhat, (3)moderately, (4) considerably, and (5)very much), hence the scale is a 5- to 15 point range. The three items are the patient's verbal report (feeling shaky, jittery, jumpy), observed behavior consistent with anxiety during the interview (e.g. appearing frightened, shaky, restless) and somatic complains (e.g., sweating, trembling, heart pounding).
  COVI Rating Scale total score is the sum of items 1 - 3.
Time Frame: 8 weeks
Population: ITT Population: Randomized and received at least one dose of the study drugs.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rufinamide | Placebo
Number analyzed (Participants) | 115 | 114
score on a scale
  Screening | 10.7 (1.39) | 10.5 (1.26)
  Baseline | 10.7 (1.35) | 10.6 (1.33)
  Week 3: number analyzed (Participants) | 102 | 101
  Week 3 | 8.3 (2.51) | 8.1 (1.99)
  Week 6: number analyzed (Participants) | 91 | 98
  Week 6 | 7.5 (2.51) | 7.6 (2.21)
  Week 8: number analyzed (Participants) | 84 | 92
  Week 8 | 7.1 (2.50) | 7.4 (2.17)
  Last Observation: number analyzed (Participants) | 109 | 110
  Last Observation | 7.7 (2.73) | 7.7 (2.29)

ADVERSE EVENTS:
Time Frame: 8 Weeks
Description: Based on the Safety/Intent-to-Treat (ITT) population. This was defined as all randomized patients who received at least one dose of study medication.
Groups:
- Placebo: 0 mg tablet
Arm/Group | Rufinamide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/114
Serious Adverse Events (participants affected / at risk) | 1/115 | 1/114
Other Adverse Events (participants affected / at risk) | 75/115 | 72/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rufinamide (N=115) | Placebo (N=114)
Acute Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Ecotopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rufinamide (N=115) | Placebo (N=114)
Vision Blurred (Eye disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 8 (8) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 4 (4)
Dry Mouth (Gastrointestinal disorders) | 6 (8) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 10 (12) | 12 (13)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (4)
Fatigue (General disorders) | 4 (4) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 9 (11)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Athralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Dizziness (Nervous system disorders) | 6 (7) | 7 (8)
Headache (Nervous system disorders) | 14 (16) | 22 (24)
Sedation (Nervous system disorders) | 3 (3) | 1 (2)
Somnolence (Nervous system disorders) | 12 (12) | 10 (10)
Anxiety (Psychiatric disorders) | 4 (4) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (4) | 4 (5)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding the study results for a period up to 30 days from the date the communication is submitted to the sponsor. The sponsor shall have the right to defer proposed publication an additional 60 days from the end of the review period. The sponsor cannot require changes to the communication and cannot unilaterally extend the embargo.